CLINICAL TRIAL: NCT02725229
Title: Comparison of Transcutaneous Electrical Nerve Stimulation and Parasternal Block for Postoperative Pain Management After Cardiac Surgery
Brief Title: Parasternal Block and TENS for Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AntalyaTRH 011
Record Dates: First submitted 2016-03-23; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Parasternal block; Sternotomy; TENS
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- parasternal block group (Active Comparator): Patients in this group will be randomized to receive an parasternal block and PCA.
  Interventions: Procedure: parasternal block
- TENS group (Active Comparator): Patients in this group will be randomized to receive an TENS and PCA.
  Interventions: Device: TENS group
- control group (Active Comparator): Patients in this group will be randomized to receive an PCA.
  Interventions: Device: control group

INTERVENTIONS:
Procedure: parasternal block — parasternal block and PCA for sternotomy pain
  Other Names: Levobupivacaine
  Arms: parasternal block group
Device: TENS group — TENS and PCA for sternotomy pain
  Other Names: TENS device
  Arms: TENS group
Device: control group — PCA for sternotomy pain
  Other Names: PCA device
  Arms: control group

SUMMARY:
the objective of the present study was to compare the efficacy of TENS and parasternal block with local anesthetic infiltration in relieving pain during the first 24 h period following median sternotomy.

DETAILED DESCRIPTION:
Patients experiencing pain after undergoing cardiac surgery may also experience prolonged immobilization, insufficient respiratory functions and the inability to cough due to median sternotomy. Invasive and noninvasive interventions such as epidural analgesia, local regional blockade and the use of intravenous (IV) opioids, are used for postoperative pain management. Transcutaneous electrical nerve stimulation (TENS) is a noninvasive technique that is effective for postoperative pain management. It has been demonstrated to produce effective analgesia and reduce postoperative opioid requirements in patients undergoing cardiac surgery, and it has no side effects. Parasternal local anesthetic infiltration around the sternum has been demonstrated to be useful in providing early postoperative analgesia, reducing opioid requirements and, therefore, producing a potential positive effect on recovery. The present prospective, randomized controlled study included 120 patients, 18 to 65 years of age, who were scheduled for elective valve repair or coronary artery bypass graft (CABG) surgery with cardiopulmonary bypass. A random number table was used to randomly allocate patients to one of three treatment groups to relieve postoperative pain during the first 24 h following median sternotomy: parasternal block group (parasternal block combined with levobupivacaine infiltration and PCA(patient controlled analgesia)); TENS group (TENS and PCA); or the control group (PCA alone).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age,
* who were scheduled for elective valve repair or coronary artery bypass graft (CABG) surgery with cardiopulmonary bypass

Exclusion Criteria:

* previous sternotomy for CABG or heart valve surgery; emergency surgery
* ejection fraction <40%
* congestive heart failure
* an allergy to amide-based local anesthetics, opioids or benzodiazepines
* inability to provide informed consent
* prolonged cardiopulmonary bypass time (>145 min)
* previous experience with TENS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-06; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scores | Assessed 24 hours after to intensive care unit admission

SECONDARY OUTCOMES:
Supplemental morphine used | Assessed 24 hours after to intensive care unit admission
Extubation time | Assessed 24 hours after to intensive care unit admission
Length of ICU stay | Assessed 24 hours after to intensive care unit admission
Length of hospital stay | Assessed 10 days after to intensive care unit admission
Supplemental tramadol used | Assessed 24 hours after to intensive care unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Kavrut Ozturk, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozturk NK, Baki ED, Kavakli AS, Sahin AS, Ayoglu RU, Karaveli A, Emmiler M, Inanoglu K, Karsli B. Comparison of Transcutaneous Electrical Nerve Stimulation and Parasternal Block for Postoperative Pain Management after Cardiac Surgery. Pain Res Manag. 2016;2016:4261949. doi: 10.1155/2016/4261949. Epub 2016 Apr 12. PMID 27445610